CLINICAL TRIAL: NCT05374967
Title: The Effect of a Multimodal Lifestyle Intervention on Chronic Fatigue in Patients With Inflammatory Bowel Disease
Acronym: Multi-IBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Medical Center Haaglanden (Other); Voeding Leeft (Unknown)
Responsible Party: Principal Investigator, Pieter Maljaars, Principal Investigator, Leiden University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL77752.058.21
Record Dates: First submitted 2022-04-07; First posted 2022-05-16 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Inflammatory Bowel Diseases; Fatigue
Keywords: IBD; Crohn's disease; Ulcerative colitis; Inflammatory Bowel Disease; Fatigue; Lifestyle
MeSH Terms: conditions — Inflammatory Bowel Diseases; Fatigue; Crohn Disease; Colitis, Ulcerative | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): The control group will receive the current standard of care: an informational brochure on how to cope with fatigue.
  Interventions: Other: Control group
- Lifestyle intervention (Experimental): Participants will undergo a multimodal lifestyle intervention, which focuses on nutrition, sleep, stress, and exercise. The lifestyle intervention includes digital lessons/webinars and online counseling by a nutritionist and a lifestyle coach.
  Interventions: Behavioral: Lifestyle intervention: Live with IBD

INTERVENTIONS:
Behavioral: Lifestyle intervention: Live with IBD — A digital lifestyle intervention divided into two phases:
  1. An intensive phase lasting six months
  2. a facultative phase lasting six months
  During the Intensive Phase, participants will receive regular counseling by a nutritionist and a lifestyle coach in groups of 25 people. Participants will also follow five online meetings focusing on either nutrition, exercise, sleep, and stress. In addition, participants will have 24/7 access to an online platform that contains additional information, challenges, recipes, and peer-support groups. Finally, during the facultative phase, participants can attend smaller group sessions for additional counseling by a nutritionist or a lifestyle coach; these sessions will be organized every six to 12 weeks.
  Other Names: Leef! met IBD
  Arms: Lifestyle intervention
Other: Control group — The standard of care for patients with IBD suffering from chronic fatigue.
  Arms: Control group

SUMMARY:
Chronic fatigue is highly prevalent in patients with conditions characterized by chronic inflammation of the gastrointestinal tract, also known as Inflammatory Bowel Disease (IBD). Chronic fatigue has multiple causes, including alterations in immune system or gut microbiota, psychological factors, and sleeping problems. Unsurprisingly, fatigue has been associated with decreased quality of life, general well-being, and work productivity. Very few patients experience resolution in fatigue, emphasizing the need for new therapies. It has been shown that lifestyle interventions can improve most of fatigue-driving factors. Hence, the investigators hypothesize that a multimodal lifestyle intervention focusing on nutrition, sleep, stress, and exercise will improve chronic fatigue in patients with IBD. During this multicenter, controlled trial, the investigators will compare a multimodal lifestyle intervention to a standard therapy (i.e., an informational brochure on how to cope with chronic fatigue).

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Established IBD diagnosis (Crohn's disease, Ulcerative colitis, or IBD-unclassified)
* Biochemical remission (fecal calprotectin ≤150 mcg/g)
* Clinically significant fatigue (visual analog score 4-8 out of 10)
* Willing and able to attend digital group sessions as a part of the intervention

Exclusion Criteria:

* Documented comorbidities such as severe cardiac failure (classified as NYHA 3-4), chronic kidney disease, myelodysplastic syndrome, Chronic Obstructive Pulmonary Disease (COPD), inherited metabolic diseases (e.g., phenylketonuria, mitochondrial or uric acid cycle pathologies), diabetes type 1
* Documented history of malignancy within the last three years before inclusion except for dermatological cancers such as basal cell carcinoma or squamous cell carcinoma
* Documented history of psychiatric diseases, eating disorders, or addiction. Exception: patients with a history of depression and/or under treatment with antidepressants; however, at inclusion the patients must have a Hospital Anxiety Depression Scale (HADS) score <11 for the depression subscale
* Documented familial hypercholesterolemia
* Diabetes type 2 treated with insulin or other medications such as sulfonylureas, glinides, alpha-glucosidase inhibitors, etc. The only exception is biguanides-metformin
* BMI <18.5 or >35 kg/m2
* Clinically significant anemia (Hb <7.0 mmol/l in females, Hb <8.0 mmol/l in males) with the exception of marginal normocytic or macrocytic anemia (MCV >100 fL and Hb >7.0 mmol/L for females and Hb >8.0 mmol/L for males) as a result of IBD-therapy related myelosuppression
* Vitamin B12 or folic acid deficiency
* Iron deficiency (defined as ferritin <30 μg/l)
* Vitamin D deficiency (<30 nmol/l)
* History of prior bariatric surgery or upper gastrointestinal surgery such as Roux-Y reconstruction or (partial) gastrectomy due to benign or malignant pathologies
* Pregnancy or active breastfeeding
* Unwillingness to follow the lifestyle program, i.e. people that do not want to eat fish, vegans
* Any change in IBD-related systemic medication within the last three months of intervention. Changes in medication dose are allowed up to 1 month before the start of the intervention. Exception: changing the route of administration (e.g., switching from intravenous infliximab to subcutaneous infliximab) or change in therapy due to side effects such as an allergic reaction or cutaneous conditions.
* Recent major surgery, e.g. laparotomy in the last four weeks
* Extended hospitalization (a >2-week admission) within four weeks before inclusion
* Unable to speak and understand Dutch language
* Participation in another study with lifestyle intervention or active consultation with a lifestyle coach on patient's initiative
* Previous participation in the IBD-tailored program by Voeding Leeft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue at six months | Six months after starting the intervention
  Percentage of patients who experience a reduction in fatigue at six months compared between the intervention and the control group. The reduction in fatigue is defined as any increase in The Functional Assessment of Chronic Illness Therapy - Fatigue ((FACIT-F) score (0-160 with lower scores indicating worse fatigue) at six months compared with the baseline.

SECONDARY OUTCOMES:
Mean change in fatigue (FACIT-F) | at three months, at 12 months after the start of the intervention.
  Mean change in fatigue (measured by FACIT-F questionnaire 0-160 with lower scores indicating worse fatigue) compared between the intervention and the control; compared at different study time points.
Mean change in fatigue (fatigue VAS) | at three months, at 12 months after the start of the intervention.
  Mean change in fatigue (measured by a fatigue visual analog scale (VAS) 0-10 with higher scores indicating worse fatigue) compared between the intervention and the control; compared at different study time points.
Mean change in quality of life (SIBDQ) | at three months, at six months, and at 12 months after the start of the intervention.
  Mean change in quality of life (measured by Short Inflammatory Bowel Disease Questionnaire (SIBDQ) 10-70 with higher scores indicating better quality of life) compared between the intervention and the control group; compared at different study time points.
Mean change in quality of life (EQ-5D VAS) | at three months, at six months, and at 12 months after the start of the intervention.
  Mean change in quality of life (measured by EuroQoL 5 Dimension Visual Analog Score (EQ-5D VAS) 0-100 with higher scores indicating better quality of life) compared between the intervention and the control group; compared at different study time points.
Mean change in activity impairment | at six months and at 12 months after the start of the intervention.
  Mean change in activity impairment (measured by Work Activity and Productivity Impairment: Inflammatory Bowel Disease (WPAI:IBD) 0-100% with higher percentages indicating greater impairment) questionnaire) compared between the intervention and the control group; compared at different study time points.
Mean Clinically Important Difference in fatigue (FACIT-F) | at three months, at six months, and at 12 months after the start of the intervention.
  Percentage of participants who reached the Mean Clinically Important Difference (MCID) in the FACIT-F (MCID = 4) scores compared between the intervention and control group at different time points.
Mean Clinically Important Difference in quality of life (SIBDQ) | at three months, at six months, and at 12 months after the start of the intervention.
  Percentage of participants who reached the Mean Clinically Important Difference (MCID) in the SIBDQ (MCID = 9) scores compared between the intervention and control group at different time points.
Mean Clinically Important Difference in quality of life (EQ-5D VAS). | at three months, at six months, and at 12 months after the start of the intervention.
  Percentage of participants who reached the Mean Clinically Important Difference (MCID) in the EQ-5D VAS (MCID = 4.2) scores compared between the intervention and control group at different time points.
Mean Clinically Important Difference in activity impairment (WPAI:IBD) | at six months and at 12 months after the start of the intervention.
  Percentage of participants who reached the Mean Clinically Important Difference (MCID) in the WPAI:IBD (MCID= 7) scores compared between the intervention and control group at different time points.
Mean change in dietary quality measured by Adjusted Mediterranean Diet Serving Score | at three months, at six months, and at 12 months after the start of the intervention.
  Mean change in dietary quality (measured by Adjusted Mediterranean Diet Serving Score (Adjusted-MDSS) 0-17 with higher scores indicating better diet quality and adherence to the diet) compared between the intervention and the control group; compared at different study time points.
Mean change in physical exercise | at three months, at six months, and at 12 months after the start of the intervention.
  Mean change in physical exercise (Short QUestionnaire to ASsess Health-enhancing physical activity (SQUASH) expressed in minutes of light/moderate/intensive exercise per week) compared between the intervention and the control group; compared at different study time points.
Mean change in perceived stress | at three months, at six months, and at 12 months after the start of the intervention.
  Mean change in perceived stress (measured by Perceived Stress Scale (PSS) 0-40 with higher scores indicating higher perceived stress) compared between the intervention and the control group; compared at different study time points.
Mean change in coping with the illness | at three months, at six months, and at 12 months after the start of the intervention.
  Mean change in coping (measured by Brief Illness Perception Questionnaire (B-IPQR) 0-10 with higher scores indicating a more threatening view of the illness) compared between the intervention and the control group; compared at different study time points.
Mean change in medical consumption | at three months, at six months, and at 12 months after the start of the intervention.
  Mean change in medical consumption (measured by iMTA Medical Consumption Questionnaire (iMCQ) expressed as incurred costs per timepoint with higher costs indicating higher medical consumption) compared between the intervention and the control group; compared at different study time points.
Mean change in sleep quality | at three months, at six months, and at 12 months after the start of the intervention.
  Mean change in sleep quality (measured by Pittsburgh Sleep Quality Index (PSQI) 0-21 with higher scores indicating worse sleep quality) compared between the intervention and the control group; compared at different study time points.
Correlation between fatigue and lifestyle (i.e., nutrition, exercise, sleep, stress) | baseline, at six months and at 12 months after the start of the intervention.
  Correlation between changes in lifestyle parameters and effect parameters (i.e., which part of the lifestyle intervention (e.g., physical activity or sleep quality) improved fatigue scores).
Correlation between locus of control and lifestyle changes | baseline, at six months and at 12 months after the start of the intervention.
  Correlation between locus of control (Health Monitor questionnaire) at baseline and changes in lifestyle parameters and effect parameters.
Cost-effectiveness of the intervention | at six months and at 12 months after the start of the intervention.
  Cost-effectiveness of the intervention based on Quality-Adjusted Life Years (QALY's) expressed as 1 (perfect health) to 0 (dead).

CONTACTS AND LOCATIONS:
Overall Officials: P.W.J. Maljaars, MD, PhD, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center (LUMC), Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391